CLINICAL TRIAL: NCT00374894
Title: The Combined Effect of 2,3-Dimercaptosuccinic Acid and Multi-Nutrients on Children in Lead Poisoning
Status: Completed | Type: Observational
Sponsor: China Medical University, China (Other)
Other Study IDs: 20032063 - 2001102049
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2006-09-12 (Estimated); Status verified 2004-04

CONDITIONS: Lead Poisoning
Keywords: 2,3-dimercaptosuccinic acid; Blood Lead Levels; children; multi-nutrients
MeSH Terms: conditions — Lead Poisoning | interventions — Succimer

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: 2,3-dimercaptosuccinic acid

SUMMARY:
Lead poisoning remains a common disease among children despite successful public health efforts that reduced its prevalence.Our study was designed to test the hypothesis that lead-poisoning children (BLLs:100-440µg/L) who were given DMSA and multi-nutrients would have a greater fall than children of other groups at 12 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Initial BLLs 100-440µg/L
* Age 3-6y
* No more than two main residences
* House cleaned (no lead contaminated)
* Normal intake history and physical

Exclusion Criteria:

* Chelation in the past 12 weeks
* Concomitant Fe deficiency(ferritin<16ng/ml)
* Hemoglobin<10.5g/dL
* Medications affecting mineral metabolism

Ages: 3 Years to 6 Years | Sex: All
Age Groups: Child
Enrollment: 500
Dates: Start 2004-03; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Jin Ya ping, professor, Study Director — Department of Environmental and Occupational Health
Locations (1):
- China Medical University, Shenyang, Liaoning, China

REFERENCES:
- [Result] CDC．Preventing lead poisoning in young children［R］. U.D.Dept of health and Human services 1991:1.